CLINICAL TRIAL: NCT06733753
Title: Ultrasound-guided Thermal Ablation for Bethesda III/IV Thyroid Nodules: A Multicenter Study
Brief Title: Ultrasound-guided Thermal Ablation for Bethesda III/IV Thyroid Nodules
Status: Recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yu-kun Luo, Clinical Professor, Chinese PLA General Hospital
Other Study IDs: 2024-656
Record Dates: First submitted 2024-12-07; First posted 2024-12-13 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ultrasound-guided thermal ablation: ultrasound-guided thermal ablation
  Interventions: Procedure: ultrasound-guided thermal ablation

INTERVENTIONS:
Procedure: ultrasound-guided thermal ablation — microwave ablation, radio frequency ablation, laser ablation

SUMMARY:
To evaluate the long-term outcomes of ultrasound-guided thermal ablation for Bethesda III/IV thyroid nodules

DETAILED DESCRIPTION:
To evaluate and predict the long-term clinical outcomes of ultrasound-guided thermal ablation for Bethesda III/IV thyroid nodules

ELIGIBILITY:
Inclusion Criteria:

1. confirmation of Bethesda III or IV on fine- needle aspiration and negative on Braf V600E test
2. no clinical or imaging evidences of extrathyroidal extension, lymph node metastasis and distant metastasis on ultrasound, neck and chest CT
3. refusal or ineligibility for surgery
4. follow-up time ≥12 months

Exclusion Criteria:

1. follicular neoplasm or malignancy findings on biopsy
2. no suspicious of malignancy in US
3. patients with contra-lateral vocal cord paralysis
4. follow- up time less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Bethesda III/IV thyroid nodules
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
volume reduction rate | through study completion, an average of 6 months
  The volume reduction rate (VRR)was calculated by the equations: VRR=([initial volume-final volume] × 100)/initial volume

SECONDARY OUTCOMES:
rate of complications | 1 week
  complications of ablation
rate of nodule regrowth | through study completion, an average of 6 months
  Regrowth was defined as ≥50% volume increase compared to the previously recorded smallest volume during the follow-up
rate of change of thyroid function | through study completion, an average of 6 months
  thyroid function test, including free triiodothyronine, free thyroxine, thyroid stimulating hormone, thyroid peroxidase antibody and anti-thyroglobulin antibodies
rate of delayed surgery | through study completion, an average of 1 year
  patients underwent surgery after ablation because of anxiety or unsatisfactory about the volume reduction
cosmetic score | through study completion, an average of 6 months
  The cosmetic score was assessed by a physician (1, no palpable mass; 2, no cosmetic problem but palpable mass; 3, a cosmetic problem on swallowing only; and 4, a readily detected cosmetic problem)
symptom score | through study completion, an average of 6 months
  The symptom score was self-measured by patients using a 10-cm visual analogue scale (grade 0-10)
rate of disappearance | through study completion, an average of 6 months
  complete disappearance of ablated nodule on ultrasound and contrast-enhanced ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Yukun Luo, Principal Investigator — Chinese PLA General Hospital
Locations (2):
- China (2):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No